CLINICAL TRIAL: NCT07064161
Title: A Double-Blind Randomized Controlled Trial on the Efficacy of Hydrocolloid Dressing vs. Topical Antibiotic on Wound Healing of Post-Punch Biopsy Wounds Among Patients in a Tertiary Hospital in Manila
Brief Title: Efficacy of Hydrocolloid Dressing vs. Topical Antibiotic on Wound Healing of Post-Punch Biopsy Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santo Tomas Hospital, Philippines (Other)
Responsible Party: Principal Investigator, Fiona Bianca V. Enriquez, Principal Investigator, University of Santo Tomas Hospital, Philippines
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-06-047-TR-AP
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Biopsy Wound
Keywords: Biopsy; Wound Healing; Bandages, Hydrocolloid; Dermatology; Anti-Bacterial Agents
MeSH Terms: interventions — Mupirocin; Pharmaceutical Preparations; Anti-Infective Agents; Bandages, Hydrocolloid; Colloids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocolloid Dressing (Experimental): Skin punch biopsy wound treated with hydrocolloid dressing.
  Interventions: Drug: Hydrocolloid Dressing (DuoDERM CGF)
- Topical Antibiotic (Experimental): Skin punch biopsy wound treated with topical antibiotic.
  Interventions: Drug: Mupirocin (drug)

INTERVENTIONS:
Drug: Mupirocin (drug) — Wounds were dressed with gauze impregnated with mupirocin ointment covered by a transparent dressing (Tegaderm)
  Other Names: Mupirocin ointment; Antimicrobial; Topical antibacterial
  Arms: Topical Antibiotic
Drug: Hydrocolloid Dressing (DuoDERM CGF) — Wounds were dressed with a 1-inch size Duoderm Control Gel Formula hydrocolloid dressing
  Other Names: hydrocolloid
  Arms: Hydrocolloid Dressing

SUMMARY:
The main objective of this study is to determine the efficacy of using hydrocolloid dressing on wound healing of post-punch biopsy wounds vs topical antibiotic. Specifically, it aims to measure the following parameters: the presence or absence of infection, the clinical estimate of reepithelialization, the clinical estimate of wound closure, scar formation, pigmentation of scar, and the cosmetic appearance of the wound.

The study is a double-blind randomized controlled trial which will be conducted at the Dermatology outpatient department and the private clinics of dermatology consultants of the University of Santo Tomas Hospital. Patients who will be included are those who are 18 to 64 years of age with clean cutaneous lesions. Excluded from this study are those who have infected wounds, those who have conditions with poor tendency to heal including diabetes mellitus, peripheral vascular disease, history of keloid formation, those currently receiving anticoagulation therapy or systemic corticosteroids, and those known to have hypersensitivity to topical antibiotics.

The primary outcome measure is the proportion of patients who achieved better overall healing when treated with hydrocolloid dressing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 to 64 years old with clean cutaneous lesions who underwent skin punch biopsy using 3-mm disposable biopsy puncher.

Exclusion Criteria:

* Patients with infected wounds.
* Patients with conditions with poor tendency to heal including diabetes mellitus, peripheral vascular disease, history of keloid formation, patients currently receiving anticoagulation therapy or systemic corticosteroids.
* Patients known to have hypersensitivity to topical antibiotics.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Absence or Presence of Infection | 5 days after punch biopsy.
  Absent - millimeters of surrounding erythema or equivocal findings Present - as inferred by indurated erythema or purulent discharge
Clinical Estimate of Reepithelialization | 5 days after punch biopsy
  Rated on a scale of:
  * 0% to 25%
  * 26% to 50%
  * 51% to 75%
  * 76% to 100%
Clinical Estimate of Wound Closure | 5 days after punch biopsy
  Rated on a scale of:
  * 0% to 25%
  * 26% to 50%
  * 51% to 75%
  * 76% to 100%
Scar Formation | 5 days after punch biopsy
  Select one of the following for the assessment:
  * Unhealed
  * Depressed or Atrophied
  * Normal fine-line scar
  * Hypertrophied scar or Keloid
Scar Pigmentation | 5 days after punch biopsy
  Select one of the following for the assessment:
  * Indeterminate or Unhealed
  * Normal
  * Hyperpigmented
  * Hypopigmented
Cosmetic Appearance | 5 days after punch biopsy
  Select one of the following for the assessment:
  * Indeterminate or Unhealed
  * Poor
  * Fair
  * Good
  * Excellent

CONTACTS AND LOCATIONS:
Locations (1):
- University of Santo Tomas Hospital, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No
Sharing of the individual participant data was not part of the patient informed consent form.

REFERENCES:
- [Background] 17. World Health Organization. Antimicrobial resistance. World Health Organization. Published November 21, 2023. https://www.who.int/news-room/fact-sheets/detail/antimicrobial-resistance
- [Background] Armstrong RB, Nichols J, Pachance J. Punch biopsy wounds treated with Monsel's solution or a collagen matrix. A comparison of healing. Arch Dermatol. 1986 May;122(5):546-9. PMID 3707170
- [Background] Holmes SP, Rivera S, Hooper PB, Slaven JE, Que SKT. Hydrocolloid dressing versus conventional wound care after dermatologic surgery. JAAD Int. 2021 Dec 21;6:37-42. doi: 10.1016/j.jdin.2021.11.002. eCollection 2022 Mar. PMID 34993497
- [Background] Li J, Chen J, Kirsner R. Pathophysiology of acute wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):9-18. doi: 10.1016/j.clindermatol.2006.09.007. PMID 17276196
- [Background] Schmitt M, Vergnes NP, Canarelli JP, Gailhrd S, Daoud S, Dodat H, Lascombes P, Melin NY, Morisson-Lacombe G, Revillon Y. Evaluation of a hydrocolloid dressing. J Wound Care. 1996 Oct 2;5(9):396-399. doi: 10.12968/jowc.1996.5.9.396. PMID 27935418
- [Background] Heffernan A, Martin AJ. A comparison of a modified form of Granuflex (Granuflex Extra Thin) and a conventional dressing in the management of lacerations, abrasions and minor operation wounds in an accident and emergency department. J Accid Emerg Med. 1994 Dec;11(4):227-30. doi: 10.1136/emj.11.4.227. PMID 7894807
- [Background] Wright A, MacKechnie DW, Paskins JR. Management of partial thickness burns with Granuflex 'E' dressings. Burns. 1993 Apr;19(2):128-30. doi: 10.1016/0305-4179(93)90034-6. PMID 8471145
- [Background] Hermans MH, Hermans RP. Preliminary report on the use of a new hydrocolloid dressing in the treatment of burns. Burns Incl Therm Inj. 1984 Dec;11(2):125-9. doi: 10.1016/0305-4179(84)90135-9. PMID 6395938
- [Background] Hulten L. Dressings for surgical wounds. Am J Surg. 1994 Jan;167(1A):42S-44S; discussion 44S-45S. doi: 10.1016/0002-9610(94)90010-8. PMID 8109684
- [Background] Michie DD, Hugill JV. Influence of occlusive and impregnated gauze dressings on incisional healing: a prospective, randomized, controlled study. Ann Plast Surg. 1994 Jan;32(1):57-64. doi: 10.1097/00000637-199401000-00011. PMID 8141537
- [Background] Estienne G, Di Bella F. [The use of DuoDerm in the surgical wound after surgical treatment of pilonidal fistulae using the open method]. Minerva Chir. 1989 Oct 15;44(19):2089-92. Italian. PMID 2616009
- [Background] Viciano V, Castera JE, Medrano J, Aguilo J, Torro J, Botella MG, Toldra N. Effect of hydrocolloid dressings on healing by second intention after excision of pilonidal sinus. Eur J Surg. 2000 Mar;166(3):229-32. doi: 10.1080/110241500750009339. PMID 10755338
- [Background] Thomas S. Hydrocolloid dressings in the management of acute wounds: a review of the literature. Int Wound J. 2008 Dec;5(5):602-13. doi: 10.1111/j.1742-481X.2008.00541.x. PMID 19134061
- [Background] Demidova-Rice TN, Hamblin MR, Herman IM. Acute and impaired wound healing: pathophysiology and current methods for drug delivery, part 1: normal and chronic wounds: biology, causes, and approaches to care. Adv Skin Wound Care. 2012 Jul;25(7):304-14. doi: 10.1097/01.ASW.0000416006.55218.d0. PMID 22713781
- [Background] Lazarus GS, Cooper DM, Knighton DR, Margolis DJ, Pecoraro RE, Rodeheaver G, Robson MC. Definitions and guidelines for assessment of wounds and evaluation of healing. Arch Dermatol. 1994 Apr;130(4):489-93. PMID 8166487
- [Background] Mendonca RJ, Coutinho-Netto J. Cellular aspects of wound healing. An Bras Dermatol. 2009 Jul;84(3):257-62. doi: 10.1590/s0365-05962009000300007. English, Portuguese. PMID 19668939
- [Background] Ramsey ML, Conrad E, Chen RL, Rostami S. Skin Biopsy. 2025 Sep 15. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470457/ PMID 29262109

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT07064161/Prot_SAP_002.pdf
  • Informed Consent Form (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT07064161/ICF_001.pdf